CLINICAL TRIAL: NCT02505581
Title: Preoperative Oral Antibiotics and Surgical Site Infections in Colon Surgery Without Mechanical Bowel Preparation. A Prospective, Multicentre, Single Blinded, Randomized Trial (ORALEV Study)
Brief Title: Parenteral Antibiotics Compared to Combination of Oral and Parenteral Antibiotics in Colorectal Surgery Prophylaxis
Acronym: ORALEV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2014-002345-21
Record Dates: First submitted 2015-06-15; First posted 2015-07-22 (Estimated); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Surgical Wound Infection
Keywords: Postoperative Wound Infection; Surgical Wound Infection; Colorectal Surgery Infection Prophylaxis
MeSH Terms: conditions — Surgical Wound Infection | interventions — Ciprofloxacin; Metronidazole; Cefuroxime

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral + Parenteral prophylaxis (Experimental)
  Interventions: Drug: Extra dosage - cefuroxime (750mg) I.V; Procedure: Colorectal Surgery; Drug: Ciprofloxacin 750 mg oral; Drug: Metronidazole 250 mg oral; Drug: Cefuroxime 1.5 g Intravenous; Drug: Metronidazole 1 g Intravenous
- Only Parenteral prophylaxis (Active Comparator)
  Interventions: Drug: Extra dosage - cefuroxime (750mg) I.V; Procedure: Colorectal Surgery; Drug: Cefuroxime 1.5 g Intravenous; Drug: Metronidazole 1 g Intravenous

INTERVENTIONS:
Drug: Extra dosage - cefuroxime (750mg) I.V — In both groups a second intravenous dose of cefuroxime (750mg) will be administered if the intraoperative time elongates more than three hours or there is an intraoperative bleeding over 1000cc
Procedure: Colorectal Surgery — Both groups undergo colorectal surgery. This section does not include rectal surgery ( see Inclusion/exclusion criteria)
Drug: Ciprofloxacin 750 mg oral — An oral antibiotic pattern of ciprofloxacin (750 mg / 12h, 2 doses) the day before surgery.
  Arms: Oral + Parenteral prophylaxis
Drug: Metronidazole 250 mg oral — An oral antibiotic pattern of metronidazole (250 / 8h, 3 doses) the day before surgery.
  Arms: Oral + Parenteral prophylaxis
Drug: Cefuroxime 1.5 g Intravenous — An intravenous antibiotic pattern of cefuroxime 1.5 g during anesthetic induction.
Drug: Metronidazole 1 g Intravenous — An intravenous antibiotic pattern of metronidazole 1 g during anesthetic induction.

SUMMARY:
Routine antibiotics for the intravenous and oral prophylaxis of colorectal surgery will be used.

Experimental group: Patients undergoing elective colorectal surgery that involves, colonic resection.

The antibiotic prophylaxis in this group will be composed of:

An oral antibiotic pattern of ciprofloxacin (750mg / 12h, 2 doses) and metronidazole (250mg / 8h, 3 doses) the day before surgery.

+

Control group: Patients undergoing elective colorectal surgery that involves, colonic resection.

The antibiotic prophylaxis in this group will be composed of:

An intravenous antibiotic pattern of cefuroxime 1g and metronidazole 1,5gr during anesthetic induction.

In both groups a second intravenous dose of cefuroxime (750mg) will be administered if the intraoperative time elongates more than three hours or there is an intraoperative bleeding over 1000cc.

There won´t be a placebo treatment. Subject compliance will be evaluated according to the usual practice in surgical care field

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting colonic pathology
* The surgery is not contraindicated
* Diagnosis of colorectal neoplasia or diverticular disease with surgical indication (stenosis, chronic constipation, recurrent infections etc ..)
* Indication of segmentary resection or total colectomy
* Patients who agree to participate voluntarily in the study and signed an informed consent.

Exclusion Criteria:

* Patients who refuse to participate in the study.
* Patients undergoing mechanical colon preparation the day before surgery.
* Patients with rectal cancer
* Patients with intra-abdominal sepsis before surgery (abscess, diverticulitis).
* Patients who received preoperative antibiotics for any reason in the two weeks prior to surgery.
* Patients with inflammatory bowel disease (ulcerative colitis, Crohn's disease and indeterminate colitis)
* Patients presenting allergy to the drugs under study.
* Patients that will not strictly follow the assigned prophylaxis regimen
* Patients undergoing urgent surgery (<24h)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 536 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2018-11-10 (Actual)

PRIMARY OUTCOMES:
Wound infection | 30 days
  Superficial, deep, body-cavity This is a Clinical measure supported by image if necessary All the morbidity problems are reported independently

SECONDARY OUTCOMES:
Hospital stay | Participants will be followed for the duration of hospital stay, an expected average of 7 days
  Hospital stay since colorectal surgery is done
Direct Adverse Drug Reactions | 24 hours since the drug is taken
  Allergic reactions Intolerance
  •This morbidity problems are reported independently as a YES/NO variable
Occlusive problems | 30 days from surgery
  Intestinal occlusion, Anastomotic stenosis, Prolonged ileus(>5days),.... Occlusive problems, Iatrogenic problems, Impaired healing ( Anastomotic leak rate , intestinal fistula , vesical fistula, peritonitis...) Bleeding problems, Cardiac complications, Nephro-urinary complications, Respiratory complications, Vascular Complications, Gastrointestinal complications, Neurological complications, Local complications...
  •This morbidity problems are reported independently as a YES/NO variable
Iatrogenic problems | 30 days after surgery
  Damage to structures such as ureters, bowel loops artery / iliac vein ....
  •This morbidity problems are reported independently as a YES/NO variable
Impaired healing | 30 days after surgery
  * This is a Clinical measure always supported by image tests.
  * This morbidity problems are reported independently as a YES/NO variable
Bleeding problems | 30 days after surgery
  Hemoperitoneum, abdominal hematoma,anastomotic bleeding ....
  •This morbidity problems are reported independently as a YES/NO variable
Cardiac complications | 30 days after surgery
  acute myocardial infarction, angor pectoris , atrial fibrillation, acute pulmonary edema
  * This is a Clinical measure supported by more specific tests if necessary.
  * This morbidity problems are reported independently as a YES/NO variable
  * Cardiologist report will be required for including this items
Nephro-urinary complications | 30 days after surgery
  Acute urinary retention, Acute renal failure, cystitis, pyelonephritis ...
  * This is a Clinical measure supported by more specific tests if necessary.
  * This morbidity problems are reported independently as a YES/NO variable
Respiratory complications | 30 days after surgery
  Pneumonia, Atelectasis, Pulmonary embolism, Respiratory distress syndrome ...
  * This is a Clinical measure always supported by image .
  * This morbidity problems are reported independently as a YES/NO variable
Vascular Complications | 30 days after surgery
  Deep venous thrombosis, phlebitis, thrombophlebitis, ...
  * This is a Clinical measure supported by more specific test if necessary .
  * This morbidity problems are reported independently as a YES/NO variable
Gastrointestinal complications | 30 days after surgery
  Liver failure, gastrointestinal bleeding, severe malnutrition, ...
  * This is a Clinical measure supported by blood test and further test if necessary
  * This morbidity problems are reported independently as a YES/NO variable
Neurological complications | 30 days after surgery
  Disorientation, cerebral vascular accident, ...
  * This is a Clinical measure.
  * This morbidity problems are reported independently as a YES/NO variable.
  * Neurologist report will be required beyond disorientation.
Local infection | 30 days after surgery
  Superficial, deep, body-cavity
  * This is a Clinical measure supported by image if necessary
  * This morbidity problems are reported independently as a YES/NO variable
Local complications | 30 days after surgery
  Hematoma, seroma, evisceration
  * This is a Clinical measure.
  * This morbidity problems are reported independently as a YES/NO variable

CONTACTS AND LOCATIONS:
Overall Officials: Eloy Espin Basany, MD PhD, Study Chair — Hospital Universitari Vall d'Hebron Research Institute
Locations (3):
- Spain (3):
  - Hospital de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital General Universitario Vall d´Hebron, Barcelona
  - Hospital Universitari de Girona Dr. Josep Trueta, Girona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Espin Basany E, Solis-Pena A, Pellino G, Kreisler E, Fraccalvieri D, Muinelo-Lorenzo M, Maseda-Diaz O, Garcia-Gonzalez JM, Santamaria-Olabarrieta M, Codina-Cazador A, Biondo S. Preoperative oral antibiotics and surgical-site infections in colon surgery (ORALEV): a multicentre, single-blind, pragmatic, randomised controlled trial. Lancet Gastroenterol Hepatol. 2020 Aug;5(8):729-738. doi: 10.1016/S2468-1253(20)30075-3. Epub 2020 Apr 21. PMID 32325012